CLINICAL TRIAL: NCT02011516
Title: A Randomized Placebo-controlled Study of Baclofen on Brain and Behavioral Outcomes in Marijuana Dependence
Brief Title: Baclofen Effects on Marijuana Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Principal Investigator, Teresa Franklin, Research Assistant Professor of Neuroscience in Psychiatry, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 818755; CURE CANN (Other: Center for the Studies of Addiction)
Record Dates: First submitted 2013-12-05; First posted 2013-12-13 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Marijuana Dependence
Keywords: Marijuana; Addiction; fMRI; Baclofen; Treatment
MeSH Terms: conditions — Marijuana Abuse; Behavior, Addictive | interventions — Baclofen; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar pill, psychosocial intervention (Placebo Comparator): twice weekly appointments with a certified clinician
  Interventions: Behavioral: Psychosocial; Drug: Placebo
- Baclofen, psychosocial intervention (Active Comparator): 20 mg. q.i.d. twice weekly appointments with a certified clinician
  Interventions: Drug: Baclofen; Behavioral: Psychosocial

INTERVENTIONS:
Drug: Baclofen
  Other Names: Kemstro; Lioresal; Liofen; Gablofen; Beklo
  Arms: Baclofen, psychosocial intervention
Behavioral: Psychosocial
Drug: Placebo
  Other Names: Sugar pill
  Arms: Sugar pill, psychosocial intervention

SUMMARY:
Studies show that certain reminders of drug use such as the sight of someone using marijuana, pictures of blunts, particular moments throughout the day, prompt marijuana users to smoke marijuana. We are measuring the brain and behavioral responses of marijuana dependent individuals to these reminders (cues) We will examine brain responses during cue exposure and determine whether these responses are associated with treatment outcome.

We are testing the hypothesis that the medication baclofen reduces brain responses during marijuana cue exposure and/or craving in marijuana dependent individuals. Baclofen is FDA-approved for other uses, but not for the treatment of marijuana dependence. Functional magnetic resonance imaging (fMRI) will be used to measure the brain's response to marijuana cues. fMRI is a painless technique that takes special pictures of the brain (or other parts of your body). It does not involve radiation or injections.

Eligible participants will have a 50% chance of receiving placebo (sugar pill) and a 50% chance of receiving baclofen. Neither the participant nor study personnel will know whether participants are receiving baclofen or placebo. Participants will also receive twice weekly psychosocial treatment with a certified clinician. Twelve weeks of treatment will be followed by a 12 week follow up.

ELIGIBILITY:
Inclusion Criteria:

* Physically healthy, as determined by a comprehensive physical examination and approval of the study physician, and mentally stable, as determined by a psychological evaluation by a licensed clinician, males or females who meet Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) criteria for marijuana dependence, ages 18-60.
* Must be able to read. [Subjects are required to be able to read because there are several self-administered measures that they must read, understand and provide written answers.]
* Females must be non-pregnant, non-lactating and either be of non-childbearing potential (i.e. sterilized via hysterectomy or bilateral tubal ligation or at least 1 year post-menopausal) or of child bearing potential but practicing a medically acceptable method of birth control. Examples of medically acceptable methods for this protocol include barrier (diaphragm or condom) with spermicide, an intrauterine device (IUD), the Nuvaring, oral contraceptives, levonorgestrel implant, hormonal injection or complete abstinence.
* Intelligence quotient of ≥ 80.
* Provide voluntary informed consent.

Exclusion Criteria:

* Participation in a clinical trial and receipt of investigational drug(s) during the previous 60 days.
* Presence of magnetically active irremovable prosthetics, plates, pins, permanent retainer, bullets, etc. (unless a radiologist confirms that it's presence is unproblematic). An x-ray may be obtained to determine eligibility given the possibility of a foreign body.
* Current use of non-removable medicated or nicotine skin patches.
* Current or prior gambling problems (assessed by subject's self-report).
* Current treatment for marijuana dependence.
* Any other current drug dependence diagnoses (except nicotine dependence).
* Any other psychiatric diagnoses. Current diagnosis/recent history (within past 6 months) of Major Depressive Disorder (MDD).
* History of head trauma or injury causing loss of consciousness, lasting more than three (3) minutes or associated with skull fracture or inter-cranial bleeding or abnormal Magnetic Resonance Imaging (MRI).
* Claustrophobia or other medical condition preventing subject from lying in the MRI for approximately one (1) hour.
* Clinically significant cardiovascular, hematologic, hepatic (liver), renal (kidney), neurological, or endocrinological abnormalities, bloodwork, and/or electrocardiogram (EKG).
* Uncontrolled diabetes or uncontrolled hypertension.
* History of psychosis, seizures, or organic brain syndrome.
* Vision problems that cannot be corrected with glasses.
* Weight exceeding 300 pounds [Imaging data acquisition is impaired with high weight individuals].
* History of stroke.

Case-by-Case:

* Human immunodeficiency virus (HIV) positive on medication for symptoms. This will be determined on an individual basis by results from the physical examination and final approval by our study physician; all results from the physical within normal range for study inclusion.
* Use of medications or natural herbs that cause sedation or affect the brain systems that are being studied. Medication use will be evaluated by our study physician on a case-by-case basis. For example, if the subject takes Benadryl but can safely refrain from use 24 hours prior to scanning sessions, they will not be excluded.
* Significant history of past alcohol or substance abuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2013-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa R Franklin, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Center for Studies of Addiction, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Timeframe: 12/2013-10/2014
  Potential subjects were recruited via word of mouth, flyers, craigslist and targeted Facebook ads
  47 potential subjects were enrolled (consented), 41 were screened, 22 passed screening, 21 baseline scan, 16 randomized, 13 treatment scan, 8 post-tx scan, 10 completed.
Pre-assignment Details: All enrolled participants, those that consented to study procedures, participated in a screening process that consisted of a physical and psychological evaluation. Those participants that did not meet our specific inclusion criteria, and/or those that met our exclusion criteria, were not assigned to groups. These individuals were given referrals.
Groups:
- Sugar Pill, Psychosocial Intervention: twice weekly appointments with a certified clinician
  Psychosocial
  Placebo
- Baclofen, Psychosocial Intervention: 20 mg. q.i.d. twice weekly appointments with a certified clinician
  Baclofen
  Psychosocial
Period: Overall Study
Arm/Group | Sugar Pill, Psychosocial Intervention | Baclofen, Psychosocial Intervention
Started | 8 | 8
Completed | 4 | 6
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill, Psychosocial Intervention | Baclofen, Psychosocial Intervention | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Urine Drug Screen
Description: Change from positive to negative over the 12 weeks of a medication regimen
Time Frame: study weeks 1-12
Measure: Count of Participants; unit: Participants
Arm/Group | Sugar Pill, Psychosocial Intervention | Baclofen, Psychosocial Intervention
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: study weeks 1-12
Arm/Group | Sugar Pill, Psychosocial Intervention | Baclofen, Psychosocial Intervention
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 4/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sugar Pill, Psychosocial Intervention (N=8) | Baclofen, Psychosocial Intervention (N=8)
Headache (General disorders) | 3 | 0
Drowsy/Sluggish (Nervous system disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Dry Mouth (General disorders) | 1 | 0
Slowed Cognition (Nervous system disorders) | 1 | 0
"High" Feeling (Nervous system disorders) | 1 | 0
Metallic Taste (Gastrointestinal disorders) | 1 | 0
Abdominal Cramping (Gastrointestinal disorders) | 0 | 1
Increase in Bowel Movements (Gastrointestinal disorders) | 0 | 1
Unintended Weight Loss (Metabolism and nutrition disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Sample size too sample to draw conclusions. No subject was able to provide a negative cannabis urine throughout treatment. A caveat is that cannabis stays in the urine for 6 weeks after final use.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes